CLINICAL TRIAL: NCT07196007
Title: Leveraging Community-clinical Linkages to Address Unmet Social Needs for People With Diabetes Living in Rural Settings
Brief Title: Leveraging Community-clinical Linkages to Address Unmet Social Needs for People With Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mary Lacy (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Mary Lacy, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 100380; 75D30124C20318 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-09

CONDITIONS: Diabetes; Diabetes Mellitus
Keywords: Unmet social needs
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: A hybrid type 2 design to evaluate the effectiveness and implementation of a community-clinic linkage (CCL) intervention in primary care clinics and a mixed methods approach to examine process factors that affect reach, acceptance, and fidelity of the CCL intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Screening Patients with Diabetes for Unmet Social Needs Plus a Community-Clinical Intervention (Experimental): The intervention will be developed by community-clinical partners and then implemented in primary care clinics in two rural communities in Kentucky. Intervention components include patient navigation using a Community Health Worker (CHW), health information technology (HIT) and quality improvement (QI) support to both clinical and community partners. Patients who screen positive for unmet social needs will work with CHWs to be connected to community organizations. The HIT support component includes implementing the Kentucky Health Information Exchange referral communication tool between clinics and community organizations and using the Kynect resource directory to refer patients to location-specific social services and community resources. The QI component includes identifying a quality improvement team and site champion, one-on-one calls with a QI advisor, action periods to test QI strategies, and support to validate health outcomes and social needs screening data.
  Interventions: Behavioral: Community-Clinical Intervention
- Usual Care (No Intervention): Clinics randomized to the control arm will receive usual care

INTERVENTIONS:
Behavioral: Community-Clinical Intervention — The intervention involves enhancing usual care for screening patients with diabetes for unmet social needs and referring those who screen positive to a Community Health Worker. Patients who screen positive for unmet social needs will work with CHWs to be connected to community organizations.
  Arms: Usual Screening Patients with Diabetes for Unmet Social Needs Plus a Community-Clinical Intervention

SUMMARY:
This study is a hybrid type 2 design to evaluate the effectiveness and implementation of a community-clinical linkage intervention in primary clinics to address unmet social needs for patients with diabetes living in rural communities. The study will take place in two rural communities in Kentucky, one in eastern Kentucky and one in western Kentucky.

DETAILED DESCRIPTION:
This study will convene clinical and community partners to complete a rapid process improvement workshop (RPIW) to co-create scalable strategies to address unmet social needs and to implement the developed strategy in primary care clinics in two rural communities in Kentucky. Results from the RPIW will be used to design an implementation template with specific implementation strategies tailored to each unique community-clinical linkage (CCL). While implementation strategies will be tailored to each CCL, the overarching intervention components for all CCL include: 1) patient navigators; 2) health information technology; and 3) quality improvement support to clinical and community partners. The finalized intervention will then be rolled out across partner clinics using a parallel-group cluster design that facilitates pragmatic randomization. The effect of the intervention on referrals will be assessed by comparing referrals between intervention and control clinics. Secondary effectiveness outcomes include status of social needs (improved or not), patient-reported quality of life, and diabetes control (A1c < 9.0% controlled vs A1c =9% uncontrolled). To evaluate implementation outcomes, we will use a mixed methods approach to examine process factors that affect reach, acceptance, and fidelity of the CCL intervention. This approach allows us to examine which strategies can be replicated and scaled up for implementation in other communities.

ELIGIBILITY:
Clinic/Staff Inclusion Criteria:

* staff at the intervention or comparison clinic

Participant Inclusion Criteria:

* age 18 or older,
* is a patient at the intervention or comparison clinic
* diagnosed with diabetes

Clinic/Staff Exclusion Criteria:

* staff not at the intervention or comparison clinic

Participant Exclusion Criteria:

* being under the age of 18,
* not a patient at the intervention or comparison clinic
* not diagnosed with diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants screened for social needs | Baseline, month 6 and month 12
  Number of participants screened for social needs intervention compared to control
Number of referrals to community based organization by primary care clinic | Baseline, month 6 and month 12
  Number of referrals to community based organization in intervention compared to control

SECONDARY OUTCOMES:
Change in Status of social needs | Baseline, month 6 and month 12
  Change in status of social needs, answered by a yes/no question as to accessed or not. Social needs include food insecurity, housing instability, difficulty with utilities, transportation issues, and intimate partner violence. Data will be reported as aggregate across needs.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) -29 | Baseline, month 6 and month 12
  The PROMIS - 29 measures health-related quality of life across seven domains. Scores are standardized on a T-score metric, with a mean of 50 and a standard deviation of 10 in a referent population. A higher score means more of the concept being measured.
Percent of participants with A1c greater than or equal to 9.0% | Baseline, month 6 and month 12
  Change in A1c level; Diabetes control (A1c < 9.0% controlled vs A1c =9% uncontrolled) via Electronic Health Record extract

CONTACTS AND LOCATIONS:
Overall Officials: Beth Lacy Leigh, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No